CLINICAL TRIAL: NCT02788760
Title: "The Length of Cervical Collar Treatment for Traumatic Sub-axial Fractures: Is Six Weeks as Safe as 12 Weeks? (A Randomized, Clinical Trial.)"
Brief Title: "The Length of Cervical Collar Treatment for Traumatic Sub-axial Fractures"
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only 32 patients included in 21 months
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Christina Høstmælingen, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/332
Record Dates: First submitted 2016-05-22; First posted 2016-06-02 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Collar Treatment of Stable Subaxial Spine Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 6 weeks (Other): This group of patients will be treated for 6 weeks with a cervical collar (Miami J collar - Össur)
  Interventions: Device: Cervical collar (Miami J collar - Össur)
- 12 weeks (Other): This group of patients will be treated for 12 weeks with a cervical collar ( (Miami J collar - Össur)
  Interventions: Device: Cervical collar (Miami J collar - Össur)

INTERVENTIONS:
Device: Cervical collar (Miami J collar - Össur) — The two groups of patients will similar in every way and will be treated with the same type of cervical collar - the only difference will be the length of treatment

SUMMARY:
Most fractures of the cervical spine are considered stable and treated with a rigid cervical collar. However no studies have to date been published addressing the length of treatment. There seems to be a significant dissimilarity between hospitals within and between countries with the length of collar treatment varying from 6 to 12 weeks. At the neurosurgical department at Oslo University Hospital, Ullevål the standard length of treatment for a stable cervical fracture is 12 weeks. This study seeks to establish whether 6 weeks of collar treatment for a specific subtype of stable fractures in the cervical spine is sufficient.

DETAILED DESCRIPTION:
The investigators will include 150 patients with a stable cervical fractures of vertebra C3-C7 with a Subaxial Cervical Spine Injury Severity (SLIC) Score 1-3 and randomize them in to two similar groups. One group will be treated with a cervical collar for 6 weeks and the other group will be treated for 12 weeks. There will be a clinical check up and a CT scan at 1, 6, 12 and 26 weeks after the initial injury. The investigators will compare the results between the two groups when it comes to fracture healing (CT based), level of function, pain and the length of sick leave with a total of 6 months of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a newly diagnosed (within 5 days of injury) fracture in vertebra C3-C7 with SLIC score 1-3
* Patients must be abel to give their consent to participate in the study

Exclusion Criteria:

* Unstable cervical fractures in need of surgery
* SLIC score >3
* Fractures of the spinous process and the transverse process in the cervical spine
* Stable fractures in in the C3-C7 vertebra combined with fractures of the C0-C2 vertebra
* Pathological fractures in the cervical spine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Fracture healing | 6 months
  The fracture healing will be assessed based on CT scans at 6 months
Visual analogue scale - neck pain and radiculopathy | 6 months
  Pain will be assessed at 6 months based on the Visual Analogue Scale and the use of pain medication will be recorded at 6 months

SECONDARY OUTCOMES:
Level of function | 6 months
  Level of function will be assessed at 6 months using the Neck Disability Index and the Karnofsky Performance Scale Index and by registering the length of sick leave at 6 months
Treatment failure | 6 months
  Treatment failure will be recorded in both arms at 6 months. Defined as the need for surgery in both groups or the need to extend the use of collar from 6 to 12 weeks in the 6 weeks group

CONTACTS AND LOCATIONS:
Overall Officials: Christina T. Høstmælingen, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Neurosurgical department, Oslo university hospital, Ullevål, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided